CLINICAL TRIAL: NCT01130584
Title: Pyruvate Kinase Isoform M2 (PKM2) as a Possible Biomarker for Cancer
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: PK01/02/10
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Cancer
Keywords: Cancer Patients
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cancer patient
  Interventions: Other: Pyruvate kinase isoform M2

INTERVENTIONS:
Other: Pyruvate kinase isoform M2

SUMMARY:
The purpose of this study is to determine if pyruvate kinase M2 (PKM2) can be used as a biomarker in cancer.

Pyruvate kinase M2 is more elevated in malignant pleural fluid than in plasma, and may be a useful biomarker to distinguish between malignant and non-malignant causes of pleural effusion. In addition, pyruvate kinase M2 has also been found to be elevated in saliva in cancer patients compared to controls. Measuring pyruvate kinase M2 in saliva may be used to diagnose cancer or monitor the treatment progress of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Any cancer patient with pleural effusion that is being drained through an indwelling chest-tube in an inpatient ward.

Exclusion Criteria:

* Patient with a pleural effusion who does not have proven cancer or whose pleural effusion is not known to be malignant.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any cancer patient
Sampling Method: Probability Sample
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Elia S, Massoud R, Guggino G, Cristino B, Cortese C, De Massimi AR, Zenobi R. Tumor type M2-pyruvate-kinase levels in pleural fluid versus plasma in cancer patients: a further tool to define the need for invasive procedures. Eur J Cardiothorac Surg. 2008 Apr;33(4):723-7. doi: 10.1016/j.ejcts.2008.01.014. Epub 2008 Feb 7. PMID 18261916
- [Background] Mazurek S. Pyruvate kinase type M2: a key regulator within the tumour metabolome and a tool for metabolic profiling of tumours. Ernst Schering Found Symp Proc. 2007;(4):99-124. doi: 10.1007/2789_2008_091. PMID 18811055